CLINICAL TRIAL: NCT07293663
Title: Comparing Mixed Reality, Video-Based, and Instructor-Led Training in Nasogastric Tube Insertion: A Randomized Controlled Trial Assessing Learning Outcomes, Usability, and Student Experiences in Nursing Education
Brief Title: Comparing Mixed Reality, Video-Based, and Instructor-Led Training for Nasogastric Tube Insertion in Nursing Students
Acronym: NURSE-TRAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: Turku University of Applied Sciences (Unknown)
Responsible Party: Principal Investigator, Marika Leppänen, Principal Investigator, University of Turku
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TY1218-RCT; TY/1218/06.01.01/2024 (Other: Ethics Committee of the University of Turku)
Record Dates: First submitted 2025-11-23; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Education, Nursing Students; Clinical Competence; Teaching Innovation; Nasogasrtic Tube Insertion; User Experience; Teaching Method
Keywords: Nasogastric Tube Insertion; Nursing Education; Mixed Reality; Video-Based Learning; Instructor-Led Training; Meta Quest 3; Nursing Clinical Skills; Randomized Controlled Trial; Nursing Students; Extended Reality in Healthcare

STUDY DESIGN:
Intervention Model Description: Participants are randomized into three parallel groups, each receiving a different instructional method for nasogastric tube (NGT) insertion training. All groups follow the same standardized protocol and instructional content. The MR group uses Meta Quest 3 mixed reality glasses with a stepwise virtual application developed in CTRL Studio. The video group watches a head-mounted smart camera recording of the procedure. The instructor-led group receives classroom-based instruction and a live demonstration. Each student performs the procedure individually on a manikin, and outcomes are assessed post-intervention and at six-month follow-up.
Who Masked: Outcomes Assessor
Masking Description: Only the outcomes assessor is blinded to group allocation. Students, instructors, and researchers are aware of the assigned intervention. The assessor evaluates NGT insertion performance without knowledge of which instructional method the student received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mixed Reality Group (Experimental): Participants in this arm receive nasogastric tube (NGT) insertion training using Meta Quest 3 mixed reality glasses. The instructional application, developed with CTRL Studio, provides stepwise virtual guidance. Students receive technical familiarization before practice. The instructional content is standardized and identical to other groups. This arm evaluates the effectiveness and usability of MR-based training.
  Interventions: Device: Mixed Reality NGT Training
- Video-Based Learning Group (Experimental): Participants in this arm receive NGT insertion training by watching a video recorded from the operator's point of view using a head-mounted, voice-controlled smart camera. The video is identical to the MR and instructor-led groups and can be replayed during practice. No verbal guidance is provided during the procedure. This arm evaluates the effectiveness and usability of video-based training.
  Interventions: Device: Video-Based NGT Training
- Instructor-Led Training Group (Control) (Experimental): Participants in this arm receive classroom-based instruction including theoretical slides and a live demonstration of the NGT insertion procedure. Students practice individually on a manikin under teacher supervision. The teacher answers questions but does not provide step-by-step coaching. This arm serves as the control condition and represents traditional teaching methods.
  Interventions: Behavioral: Instructor-Led NGT Training

INTERVENTIONS:
Device: Mixed Reality NGT Training — Participants use Meta Quest 3 mixed reality glasses with a stepwise instructional application developed in CTRL Studio. The application provides interactive virtual guidance for nasogastric tube (NGT) insertion. Students receive technical familiarization before practice. Content is standardized and identical to other groups.
  Other Names: Meta Quest 3 MR Training
  Arms: Mixed Reality Group
Device: Video-Based NGT Training — Participants watch a video of the NGT insertion procedure recorded from the operator's point of view using a head-mounted, voice-controlled smart camera. The video is identical to the MR and instructor-led groups and can be replayed during practice. No verbal guidance is provided during the procedure.
  Other Names: Video-Based Skill Training
  Arms: Video-Based Learning Group
Behavioral: Instructor-Led NGT Training — Participants receive classroom-based instruction including theoretical slides and a live demonstration of the NGT insertion procedure. Students practice individually on a manikin under teacher supervision. The teacher answers questions but does not provide step-by-step coaching.
  Other Names: Traditional Teaching; Classroom-Based Instruction; Teacher-Guided Training
  Arms: Instructor-Led Training Group (Control)

SUMMARY:
This study explores how nursing students learn to insert a nasogastric tube (NGT), a common but potentially risky clinical procedure. The goal is to compare three different teaching methods:

Mixed Reality (MR) glasses with virtual instructions Video-based learning Traditional instructor-led training

The study investigates which method leads to better learning outcomes, how usable the technologies are, and how students experience MR in their learning.

Participants will be first-year nursing students with no prior experience in NGT insertion. They will be randomly assigned to one of the three training methods, complete the procedure, and answer questionnaires about their performance and experience. Six months later, they will repeat the procedure to assess long-term learning.

DETAILED DESCRIPTION:
This randomized controlled trial investigates the effectiveness of three teaching methods Mixed Reality (MR), Video-Based Learning (VBL), and Instructor-Led Training in teaching nasogastric tube (NGT) insertion to first-year nursing students. The study aims to compare learning outcomes, usability, and user experience across these methods, and to assess long-term retention of clinical skills.

NGT insertion is a routine but high-risk procedure in nursing. Incorrect placement can lead to serious complications such as aspiration, nasal trauma, or increased mortality. Effective training is essential to ensure safe and competent practice.

Participants will be randomized into three parallel groups with identical instructional content based on a standardized NGT insertion protocol:

Mixed Reality (MR) Group (N=60) Students use Meta Quest 3 mixed reality glasses running a stepwise instructional application developed with CTRL Studio.

The MR application provides interactive, virtual guidance for each step of the NGT insertion procedure.

Prior to practice, students receive technical familiarization, including hands-on use of the MR device and navigation of the virtual interface.

The virtual content is identical to the other groups and can be replayed during practice.

Video-Assisted Group (N=60) Students watch a video of the NGT insertion procedure recorded from the operator's point of view using a head-mounted, voice-controlled smart camera.

The video content is identical to the MR and instructor-led sessions and can be replayed during practice. No additional verbal guidance is provided during practice.

Instructor-Led Group (Control) (N=60) Students receive classroom-based instruction including theoretical slides and a live demonstration of the NGT insertion procedure.

Students practice individually on a manikin under teacher supervision. The teacher answers questions but does not provide step-by-step coaching.

All students complete a pre-test on NGT theory and a demographic questionnaire. Each student performs the NGT insertion individually on a manikin during the practice phase.

After practice, students complete:

NASA-TLX workload assessment and NGT theory post-test (all groups) System Usability Scale (SUS) and User Experience Questionnaire (UEQ) (MR and video groups only) MR group also submits a written reflection on device usability.

Finally, students repeat the NGT insertion in a separate room without guidance. Performance is assessed by a blinded research assistant using a standardized NGT checklist.

The study follows the Medical Research Council (MRC) Framework for developing and evaluating complex interventions. The intervention materials are evidence-based and piloted with teachers and students before implementation. The sample size is calculated to ensure statistical power, and data will be analyzed using SPSS software. ANOVA and t-tests will be used to compare group outcomes, and qualitative data from student reflections will be analyzed using content analysis.

This study contributes to the development of evidence-based teaching strategies in nursing education. It explores how immersive technologies like MR can enhance skill acquisition, motivation, and satisfaction. The findings will inform future curriculum design and support the integration of digital tools in clinical training.

Ethical approval has been obtained, and all participants will provide informed consent. Data will be anonymized and securely stored. The study is conducted in collaboration with the University of Turku and Turku University of Applied Sciences.

ELIGIBILITY:
Inclusion Criteria:

* First-year nursing student
* Performing nasogastric tube (NGT) insertion for the first time
* No prior theoretical education or pre-material on NGT insertion procedure

Exclusion Criteria:

* Previous nursing education (e.g., practical nurse qualification)
* Diagnosis of epilepsy
* Presence of a pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
NGT Checklist Performance Score | Immediately after training; 6 months after training
  Student performance in nasogastric tube (NGT) insertion is assessed using a structured NGT checklist. Total score on the NGT checklist is 38 point. Higher scores indicate better procedural performance. The checklist evaluates both technical and non-technical procedural steps to determine clinical competence. Assessment is conducted immediately after the intervention (M1) and again six months later (M2) without instructional support.
  Checklist completed by a research assistant or staff member observing the student performing the NGT procedure on a manikin.
  The NGT checklist is based on validated tools (e.g., Kebede et al., 2024) and is designed to objectively measure students' ability to perform NGT insertion safely and correctly.

SECONDARY OUTCOMES:
User Experience Questionnaire (UEQ) | Immediately after intervention
  Students complete the User Experience Questionnaire (UEQ) after performing the NGT insertion procedure. The UEQ measures six dimensions of user experience: attractiveness, perspicuity, efficiency, dependability, stimulation, and novelty. Each dimension is scored from -3 to +3, with higher scores indicating a more positive experience. The questionnaire is used to evaluate the perceived quality and usability of the Mixed Reality and Video-Based Learning environments.
System Usability Scale (SUS) | Immediately after intervention
  Students complete the SUS questionnaire after performing the NGT procedure. The SUS is a standardized 10-item Likert-scale tool that measures perceived usability of the Mixed Reality and Video-Based Learning environments. Scores range from 0 to 100, with higher scores indicating better perceived usability.
NASA Task Load Index (NASA TLX) | Immediately after intervention
  NASA Task Load Index (NASA TLX), a multidimensional workload assessment tool. Scores range from 0 to 100, with higher scores indicating greater cognitive workload Students complete the NASA TLX questionnaire to assess cognitive workload during the NGT procedure. The tool includes six dimensions: mental demand, physical demand, temporal demand, performance, effort, and frustration.
Student Reflection Texts | Immediately after intervention
  Students who used MR glasses submit written reflections describing their learning experience, including factors that facilitated or hindered skill acquisition.
Nasogastric Tube (NGT) theory pre- and post-test | Baseline; Immediately after intervention
  Students complete a Nasogastric Tube (NGT) theory pre-test before the intervention and a post-test immediately after performing the NGT insertion procedure. Both tests use the same set of 15 questions to assess theoretical knowledge of nasogastric tube insertion. The pre-test is used to establish baseline knowledge and group homogeneity, while the post-test measures knowledge acquisition following the assigned learning method. Scores range from 0 to 15, with higher scores indicating better theoretical knowledge of NGT insertion.

CONTACTS AND LOCATIONS:
Overall Officials: Marika Leppänen, Doctoral Researcher, Principal Investigator — University of Turku, Department of Nursing Science; Heli Virtanen, Professor, Study Chair — University of Turku, Department of Nursing Science; Minna Kyttälä, Professor, Study Chair — University of Turku, Department of Education; Teijo Lehtonen, Doctor of Science (Technology), Study Chair — University of Turku, Department of Computing
Locations (1):
- Turku University of Applied Sciences, Turku, Finland

IPD SHARING:
Plan to Share IPD: No
No, individual participant data (IPD) will not be shared. The data collected in this study will be used solely for statistical analysis and the publication of aggregated results in peer-reviewed scientific articles. Due to ethical considerations, including participant confidentiality and the nature of the consent obtained, individual-level data will not be made publicly available.

DOCUMENTS (1):
  • Study Protocol (2025-12-06): https://cdn.clinicaltrials.gov/large-docs/63/NCT07293663/Prot_000.pdf